CLINICAL TRIAL: NCT05793411
Title: Risk Behaviors in Adolescents With Chronic Diseases
Acronym: Carmac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210802
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Disease; Somatic Disorders
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire risk behaviors in adolescents with chronic diseases — Questionnaire risk behaviors in adolescents with chronic diseases

SUMMARY:
Little is known about the prevalence of risk behaviors (RBs), in adolescents living with a chronic condition (CC) Objectives Main objective: To characterize the engagement of adolescents with somatic CC recognized as ALD (SCC-ALD) into RBs, compared to the French GP Secondary objectives

* To identify factors associated with RBs in adolescents with somatic CC-ALD
* To elicit strategies of preventive action of RBs in adolescents with somatic CC-ALD Methods multicenter, cross-sectional survey , based on a mixed qualitative-quantitative approach with an explanatory sequential design (2 consecutive steps): STEP 1 : QUANTITATIVE COMPONENT

  * N expected =500
  * Inclusion criteria : 14 to 18 years, With a SCC-ALD,Without cognitive impairment and/or psychiatric disease
  * Pseudonymised self-administered paper questionnaire (50 items) completed by eligible adolescents during a visit at referring hospital
  * statistical analysis : Comparative to the French GP: matching with two datasets (Enclass-HBSC 2022 and Portraits d'Adolescents 2013 surveys); identification of risk factors and risk subgroups STEP 2 : QUALITATIVE COMPONENT: Focus groups of adolescents with somatic CC-ALD (5 focus groups of 6-8 adolescents, conducted by a researcher in SHS) Perspectives

CARMAC will :

* Provide a better understanding of RBs in adolescents with severe somatic CC and
* Help develop strategies to prevent RBs to enhance the strategies of reducing the addictions to psychoactive substances and health inequalities in this population
* Serve as a methodological model for future studies

DETAILED DESCRIPTION:
Little is known about the prevalence of risk behaviors (RBs), in adolescents living with a chronic condition (CC) Objectives Main objective: To characterize the engagement of adolescents with somatic CC recognized as ALD (SCC-ALD) into RBs, compared to the French GP Secondary objectives

* To identify factors associated with RBs in adolescents with somatic CC-ALD
* To elicit strategies of preventive action of RBs in adolescents with somatic CC-ALD Methods multicenter, cross-sectional survey , based on a mixed qualitative-quantitative approach with an explanatory sequential design (2 consecutive steps) STEP 1 : QUANTITATIVE COMPONENT

  * N expected =500
  * Inclusion criteria : 14 to 18 years, With a SCC-ALD,Without cognitive impairment and/or psychiatric disease
  * Pseudonymised self-administered paper questionnaire (50 items) completed by eligible adolescents during a visit at referring hospital
  * statistical analysis : Comparative to the French GP: matching with two datasets (Enclass-HBSC 2022 and Portraits d'Adolescents 2013 surveys); identification of risk factors and risk subgroups STEP 2 : QUALITATIVE COMPONENT: Focus groups of adolescents with somatic CC-ALD (5 focus groups of 6-8 adolescents, conducted by a researcher in SHS) Perspectives

CARMAC will :

* Provide a better understanding of RBs in adolescents with severe somatic CC and
* Help develop strategies to prevent RBs to enhance the strategies of reducing the addictions to psychoactive substances and health inequalities in this population
* Serve as a methodological model for future studies

ELIGIBILITY:
Inclusion Criteria:

* 14 to 18 years, living with a somatic chronic condition, recognized as an ALD (long duration disease)

Exclusion Criteria:

* cognitive impairment and/or psychiatric disease

Ages: 14 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents living with a severe chronic condition
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of risky behaviors in adolescents with somatic chronic conditions recognized as ALD (SCC-ALD) compared to the French General Population | 6 months
  prevalence of tobacco, cannabis and alcohol us, of risky sexuality, of dangerous games

SECONDARY OUTCOMES:
Factors associated with high prevalence of risky behaviors in of adolescents with somatic chronic conditions recognized as ALD (SCC-ALD) compared to the French General Population | 6 months
  gender, age, social background, self-esteem, type of chronic condition, perceived burden of chronic condition (pain, treatment, social impact)

CONTACTS AND LOCATIONS:
Overall Officials: Helene MELLERIO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No